CLINICAL TRIAL: NCT03302845
Title: A Phase 1, Open-label, Parallel Group, Drug-drug Pharmacokinetic Interaction Study to Evaluate the Effects of Multiple-dose Omeprazole and Famotidine on the Absorption of Single-dose Telotristat Ethyl in Healthy Male and Female Subjects
Brief Title: A Phase 1 Study to Evaluate the Effects of Omeprazole and Famotidine on the Absorption of Telotristat Ethyl in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LX1606.1-110-NRM; LX1606.110 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Drug-drug Interaction
MeSH Terms: interventions — Omeprazole; Famotidine; telotristat ethyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omeprazole (Experimental): Subjects will receive one 40 mg omeprazole capsule per day for 4 days and one 250 mg telotristat ethyl tablet on two separate occasions.
  Interventions: Drug: Omeprazole 40 MG; Drug: Telotristat ethyl 250 mg
- Famotidine (Experimental): Subjects will receive one 40 mg famotidine tablet given twice daily for 4 days and one 250 mg telotristat ethyl tablet on two separate occasions.
  Interventions: Drug: Famotidine 40 mg; Drug: Telotristat ethyl 250 mg

INTERVENTIONS:
Drug: Omeprazole 40 MG — Omeprazole 40 mg capsule
  Arms: Omeprazole
Drug: Famotidine 40 mg — Famotidine 40 mg tablet
  Arms: Famotidine
Drug: Telotristat ethyl 250 mg — Telotristat ethyl 250 mg tablet

SUMMARY:
This drug-drug interaction study will evaluate the impact of two different acid reducing agents (from two different drug classes) co-administered with a single dose of telotristat ethyl.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females ≥18 to ≤ 65 years of age at the time of Screening:

  1. Females of non-childbearing potential are to be surgically sterile (documented hysterectomy, tubal ligation, or bilateral salpingo-oophorectomy) or postmenopausal (defined as at least 12 months of spontaneous amenorrhea). Females of childbearing potential must agree to use an adequate method of contraception during the study from CRU admission through Safety Follow-up. Adequate methods of contraception for subjects or partner include condom, diaphragm, or cervical cap used in conjunction with spermicidal gel, foam, cream, film, or suppository. Hormonal contraception is NOT acceptable in this study. If necessary, follicle-stimulating hormone (FSH) results >40 IU/L at Screening are confirmatory in the absence of a clear postmenopausal history.
  2. Nonsterile male subjects with sexual partners of childbearing potential must agree to use adequate methods of contraception from CRU admission through Safety Follow-up. Adequate methods of contraception for subjects or partner include the following: condom with spermicidal gel, diaphragm with spermicidal gel, coil (intrauterine device), surgical sterilization, vasectomy, oral contraceptive pill, depo-progesterone injections, progesterone implant (ie, Implanon®), NuvaRing®, Ortho Evra®; if a subject is not sexually active, but becomes active, he or his partner should use medically accepted forms of contraception.
* Body mass index ≥18.0 to ≤32.0 kg/m2 at Screening and Baseline/predose Day 1
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Able to comprehend and willing to sign an informed consent form (ICF)
* All laboratory values at Screening and CRU admission fall within normal range or are evaluated as not clinically significant (NCS) by the Investigator if outside normal range.
* Has no clinically meaningful abnormal findings during Screening and CRU admission physical examination, Screening and Baseline ECG, or Screening and Baseline vital signs
* Has the ability to understand and communicate the requirements of the study and is willing to comply with all study procedures
* Has not consumed and agrees to abstain from taking any dietary supplements, herbal products (eg, St. John's wort, garlic, or milk thistle), over-the-counter medications (OTC), supratherapeutic doses of vitamins, or prescription drugs (except as authorized by the Investigator AND Medical Monitor) from 14 days prior to CRU admission through the Safety Follow-up Visit
* Has not consumed alcohol-containing beverages for 3 days prior to CRU admission (as confirmed by alcohol breath analyzer) and agrees not to consume alcohol through the Safety Follow-up Visit
* Has not used tobacco- and/or nicotine-containing products within 60 days prior to the CRU admission and agrees to abstain from using tobacco- and/or nicotine-containing products, including e-cigarettes, through the Safety Follow-up Visit

Exclusion Criteria:

* History of any clinically significant psychiatric, renal, hepatic, pancreatic, cardiovascular, neurological, endocrinologic, hematological, or gastrointestinal (GI) abnormality
* Participation in another investigational study within 30 days of CRU admission
* Receipt of any protein- or antibody-based therapeutic agents (eg, growth hormones or monoclonal antibodies) within 3 months prior to Screening. Note: Influenza vaccine will be allowed if administered >21 days prior to CRU admission.
* Prior exposure to TE
* History of any serious adverse reaction or hypersensitivity to any inactive component of TE (ie, microcrystalline cellulose, croscarmellose sodium [disintegrant], talc, silicone dioxide, and magnesium stearate [non-bovine]), unless reaction is deemed irrelevant to the study by the Investigator and Sponsor
* History of malabsorption, bariatric surgery, gastric surgery, cholecystectomy, short-bowel syndrome, or GI surgery that may induce malabsorption
* History of any serious adverse reaction or hypersensitivity to any component of OMP or FTE
* History of any active infection within 14 days prior to first drug administration, if deemed clinically significant by the Investigator and/or Sponsor
* Positive hepatitis panel (including hepatitis B surface antigen and hepatitis C virus antibody) or positive human immunodeficiency virus antibody screens
* Existence of any surgical or medical condition that, in the judgment of the Investigator, might interfere with the absorption, distribution, metabolism, or excretion of TE (appendectomy and hernia repair are acceptable)
* Concurrent conditions that could interfere with safety and/or tolerability measurements
* Subject has donated plasma within 7 days of first drug administration.
* Subject has donated 1 or more pints of blood (or equivalent blood loss) within 30 days prior to first drug administration.
* Women who are breastfeeding or are planning to become pregnant during the study
* eGFR ≤ 89 ml/min/1.73 m2
* Positive pregnancy test (females only)
* Positive urine screen for selected drugs of abuse and cotinine at Screening or CRU admission
* Consumption of caffeine- and/or xanthine-containing products (cola, coffee, tea, chocolate, etc.) within 72 hours prior to CRU admission (Day 0) and throughout the study
* Consumption of grapefruit, Seville oranges, and grapefruit- or Seville orange-containing products within 72 hours prior to CRU admission (Day 0) and throughout the study
* Need for dietary restrictions, unless the restrictions are approved by the Investigator and Sponsor
* Inability or difficulty swallowing whole tablets
* Poor venous access as defined by the Investigator or a designee
* Any other condition that compromises the ability of the subject to provide informed consent or to comply with the objectives and procedures of this protocol, as judged by the Investigator or medical monitor
* Unable or unwilling to communicate or cooperate with the Investigator for any reason
* Employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members of the employees or the Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration of telotristat ethyl | 7 days
  Maximum observed concentration of telotristat ethyl
Time of maximum observed concentration of telotristat ethyl | 7 days
  Time of maximum observed concentration of telotristat ethyl
Area under the plasma concentration-time curve beginning from the first dose until the last quantifiable concentration of telotristat ethyl | 7 days
  Area under the plasma concentration-time curve beginning from the first dose until the last quantifiable concentration of telotristat ethyl

SECONDARY OUTCOMES:
Number of adverse events | Up to 13 days
  Number of adverse events throughout the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Covance Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided